CLINICAL TRIAL: NCT03749083
Title: A Study of the Role of Circulating Tumor DNA in Predicting the Likelihood of Organ Preservation After Clinical Complete Response to Neoadjuvant Therapy for Rectal Cancer
Status: Withdrawn | Type: Observational
Why Stopped: Funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Clinical Genomics (Unknown)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 18-304
Record Dates: First submitted 2018-11-15; First posted 2018-11-21 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Gastrointestinal Malignancies
Keywords: Gastrointestinal Malignancies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumor Sequencing: * Quality of life assessments will be collected using The Functional Assessment of Cancer Therapy- Colorectal
  * Blood for circulating tumor DNA will be collected
  Interventions: Other: The Functional Assessment of Cancer Therapy- Colorectal

INTERVENTIONS:
Other: The Functional Assessment of Cancer Therapy- Colorectal — The Functional Assessment of Cancer Therapy- Colorectal (FACT-C) questionnaire measures health-related quality of life for people with chronic illnesses.

SUMMARY:
In this research study, the investigators are looking to see if the circulating tumor DNA (genetic material), also known as ctDNA, in the blood will help them predict whether the participant's cancer will come back.

DETAILED DESCRIPTION:
In this research study, the investigator are performing blood draws to see if the presence or absence of circulating tumor DNA (ctDNA), the genetic material in the participant's cancer's cells, will help the investigators predict whether the participant's cancer will come back or not.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have achieved a clinical complete response (cCR) within 3 months of last therapy - defined as absence of residual ulceration, mass or mucosal irregularity at endoscopic assessment - following neoadjuvant therapy with chemoradiation or chemotherapy followed by radiation for stage I, II, or III non-metastatic rectal cancer. (Whitening of the mucosa with presence of telangiectasia will be accepted as cCR.)
* Participants must have original tumor tissue (formalin-fixed, paraffin-embedded specimens) available for analysis
* Participants must be 18 years of age or older.
* Participants must be able to understand and willing to sign a written informed consent document.
* Participants must have received long course chemoradiation to 40-54 Gy.
* Participants must have received at least 4 cycles of FOLFOX
* Participant must be no more than 3 months past the conclusion of initial chemoradiation of rectal cancer (i.e., end of chemoradiation).

Exclusion Criteria:

* Participants may not have any other organ cancer evident at the time of enrollment.
* Participants may not have any other concurrent serious illness that makes participation on this study impractical or clinically inappropriate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This prospective, observational, non-interventional study will enroll patients who have achieved a clinical complete response after treatment for rectal cancer and are undergoing standard surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-12-31 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
One year local recurrence rate in participants that test positive for ctDNA compared to participants that tested negative for ctDNA | 1 year
  Local recurrence will be defined as recurrence of the pathologically confirmed adenocarcinoma. This may be detected by endoscopy for intraluminal recurrence or after radical surgery for radiographic evidence of extraluminal/mesorectal recurrence. The recurrence must be in the peri-anastomic site or rectal stump, or pre-sacral area. Regional nodal recurrence and lateral pelvic lymph node recurrence of rectal cancer are also included in this definition.

SECONDARY OUTCOMES:
Local recurrence rate at any time up to 5 years in patients who have achieved a clinical complete response after rectal cancer treatment but who test positive for circulating tumor DNA at study entry | 5 years
  Local recurrence will be defined as recurrence of the pathologically confirmed adenocarcinoma. This may be detected by endoscopy for intraluminal recurrence or after radical surgery for radiographic evidence of extraluminal/mesorectal recurrence. The recurrence must be in the peri-anastomic site or rectal stump, or pre-sacral area. Regional nodal recurrence and lateral pelvic lymph node recurrence of rectal cancer are also included in this definition.
Overall rate of local recurrence by stratified KRAS/BRAF status and possibly other gene targets | 5 years
  Local recurrence will be defined as recurrence of the pathologically confirmed adenocarcinoma. This may be detected by endoscopy for intraluminal recurrence or after radical surgery for radiographic evidence of extraluminal/mesorectal recurrence. The recurrence must be in the peri-anastomic site or rectal stump, or pre-sacral area. Regional nodal recurrence and lateral pelvic lymph node recurrence of rectal cancer are also included in this definition.
Median EORTC QLQ-CR29 Score | Baseline, 6 months, 12 months, 24 months
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) for Colorectal cancer(CR) 29 item questionnaire. The survey will be given at baseline, 6, 12, and 24 months. Results will be reported as the median score for each question. A score of 1 represents 'Not at All' and 4 represents 'Very Much'.
Median SF-12 Health Survey Score | Baseline, 6 months, 12 months, 24 months
  The SF-12 is a 12 item validated questionnaire that assesses a participants view of their health. Scores will be normalized on a 100 point scale with higher scores representing better health.
Median LARS Score | Baseline, 6 months, 12 months, 24 months
  The Low Anterior Resection Syndrome (LARS) Score is used to assess bowel dysfunction. The survey is assessed on a scale of 0-42 points, with a higher score indicating worse bowel dysfunction.
Median FIQOL Score | Baseline, 6 months, 12 months, 24 months
  Fecal Incontinence Quality of Life (FIQOL) Score. Lower scores represent lower functional status.
Median Fecal Incontinence Severity Index (FISI) score | Baseline, 6 months, 12 months, 24 months
  The FISI measures incontinence for gas, mucus, liquid stool,and solid stool. The survey assesses the number of times per day that the participant experiences incontinence for gas, mucus, liquid stool,and solid stool. Higher scores represent a higher degree of fecal incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women Hospital, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: No